CLINICAL TRIAL: NCT00087256
Title: Celecoxib Polyp Prevention Trial in Participants With Resected Stage I Colon Cancer
Brief Title: Celecoxib in Preventing Polyps in Patients Who Have Undergone Surgery for Stage I Colon Cancer
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: For scientific, logistic, and administrative reasons.
Sponsor: NSABP Foundation Inc (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: NSABP P-3; NSABP-P-3
Record Dates: First submitted 2004-07-08; First posted 2004-07-12 (Estimated); Last update posted 2013-01-07 (Estimated); Status verified 2013-01

CONDITIONS: Colorectal Cancer
Keywords: stage I colon cancer; adenocarcinoma of the colon
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms | interventions — Celecoxib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1: placebo (Placebo Comparator): one placebo capsule taken orally twice a day for 3 years
  Interventions: Drug: Celecoxib
- Arm 2: celecoxib (Experimental): one 400 mg capsule taken orally twice a day for 3 years
  Interventions: Other: placebo

INTERVENTIONS:
Drug: Celecoxib
  Other Names: Celebrex
  Arms: Arm 1: placebo
Other: placebo
  Arms: Arm 2: celecoxib

SUMMARY:
RATIONALE: Chemoprevention therapy is the use of certain drugs to try to prevent the development of cancer. It is not yet known whether celecoxib is effective in preventing polyps in patients with colon cancer.

PURPOSE: Randomized phase III trial to study the effectiveness of celecoxib in preventing the development of polyps in patients who have undergone surgery for stage I colon cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare celecoxib vs placebo, in terms of decreasing the incidence of adenomatous polyps of the colon and rectum, in patients with resected stage I adenocarcinoma of the colon.

Secondary

* Compare disease-free survival of patients treated with these regimens.
* Compare the effect of these regimens on self-reported symptoms and health-related quality of life of these patients.
* Compare the quality of life of patients treated with these regimens.
* Compare the benefits of celecoxib in patients with primary tumors or polyps that express cyclo-oxygenase-2 (COX-2) with those that do not express COX-2.
* Compare the expression of signaling targets such as serine/threonine AKT, extracellular signal-regulated kinase 2 (ERK2), and endoplasmic reticulum Ca+2- ATPases in the index tumor and polyps.
* Determine the toxicity and safety of celecoxib in these patients.

OUTLINE: This is a randomized, double-blind, placebo-controlled, multicenter study. Patients are stratified according to gender, tumor stage (T1 vs T2), age (≤ 49 vs 50 to 59 vs ≥ 60 years), and current aspirin use (yes vs no). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive oral celecoxib twice daily for 3 years.
* Arm II: Patients receive oral placebo twice daily for 3 years. In both arms, treatment continues in the absence of unacceptable toxicity or the diagnosis of invasive colon cancer, carcinoma in situ of the colon or rectum, or a non-colon primary cancer.

Quality of life is assessed at baseline and then at 6, 12, 24, 36, and 42 months.

Patients are followed at 6 months and at 2 years.

PROJECTED ACCRUAL: A total of 1,200 patients (600 per treatment arm) will be accrued for this study within 2.5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the colon

  * Stage I disease
  * Distal border of tumor ≥ 12 cm from the anal verge
* Tumor completely resected within the past 90 days
* Must have undergone a preoperative or postoperative colonoscopy to the cecum (or small bowel anastomosis) within the past 90 days

  * All observed polyps must have been removed
* Patients with a history suggestive of hereditary non-polyposis colorectal cancer (HNPCC) must have a normal microsatellite instability status by immunohistochemistry or polymerase chain reaction

  * Patients with family history of colon cancer who have not been diagnosed with HNPCC are eligible
* No prior familial adenomatous polyposis
* No prior invasive cancer or carcinoma in situ of the colon or rectum
* No clinical or radiologic evidence of metastatic disease

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Zubrod 0-1

Life expectancy

* At least 10 years

Hematopoietic

* Complete blood count normal
* Platelet count normal

Hepatic

* Aspartate aminotransferase (AST) normal
* Bilirubin normal
* Alkaline phosphatase normal

Renal

* Creatinine normal

Cardiovascular

* No active ischemic heart disease
* No New York Heart Association class III or IV heart disease
* No myocardial infarction within the past 6 months
* No symptomatic arrhythmia
* No symptomatic peripheral vascular disease or carotid disease that would preclude study participation

Pulmonary

* No aspirin-sensitive asthma

Gastrointestinal

* No history of inflammatory bowel disease
* No history of upper gastrointestinal bleeding
* No history of duodenal or gastric ulcer

Other

* No known hypersensitivity to any COX-2 inhibitor, NSAIDs, aspirin, or sulfonamides
* No non-colorectal malignancy within the past 5 years except carcinoma in situ of the cervix, melanoma in situ, or basal cell or squamous cell skin cancer
* No other disease that would preclude study participation
* No psychiatric disorders, including history of clinical depression or addictive disorders, that would preclude giving informed consent or long-term compliance
* No rheumatologic or skeletal disorders requiring chronic NSAIDs or steroid therapy
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Not specified

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* See Disease Characteristics

Other

* No other concurrent investigational agents for colon cancer
* No concurrent chronic use of other cyclo-oxygenase-2 (COX-2) inhibitors, non-steroidal anti-inflammatory drugs (NSAIDs), or salicylates (e.g., aspirin)

  * Chronic use is defined as use for more than an average of 3 days per month

    * Concurrent NSAIDs allowed for up to 10 consecutive days for temporary relief due to inflammatory syndromes, injury, or postoperative pain
  * Cardioprotective doses of aspirin (≤ 81 mg/day or 325 mg every other day) allowed
* No concurrent fluconazole or lithium

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2004-07; Primary Completion 2006-04 (Actual); Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
To determine whether celecoxib 400 mg bid for 3 years will decrease the incidence of adenomatous polyps of the colon and rectum in participants with Stage I adenocarcinoma of the colon. | 60 months

SECONDARY OUTCOMES:
To access whether celecoxib will increase disease-free survival. | 60 months
To access whether celecoxib therapy affects self-reported symptoms and health-related quality of life. | 60 months
To describe the quality of life in early stage colon cancer patients. | 42 months
To evaluate if the benefits from celecoxib are more pronounced in a cohort of participants whose primary colon tumors and polyps express COX-2. | 60 months
To examine the expression of signaling targets such as serine/threonine kinase (AKT) extracellular signal-regulated kinase (ERK2), and endoplasmic reticulum Ca2+-ATPases in the index tumor and polyps. | 60 months
To monitor the toxicity and safety of celecoxib in this population. | 60 months

CONTACTS AND LOCATIONS:
Overall Officials: Norman Wolmark, MD, Principal Investigator — NSABP Foundation Inc
Locations (1):
- Allegheny General Hospital, Pittsburgh, Pennsylvania, United States